CLINICAL TRIAL: NCT07380308
Title: " Development of Primary Cultures of Diaphragmatic Myoblasts for Basic Research Purposes "
Acronym: MYODiaph
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other); UMR INSERM 1124 (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP250977; 2024-A02556-41 (Other: Ministry of Health - France)
Record Dates: First submitted 2026-01-14; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
Keywords: Diaphragmatic endometriosis; Surgical nodules resection
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Diaphragmatic samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with endometriosis requiring surgical nodules resection in the diaphragm.
  Interventions: Other: During the surgery planned as part of the routine care of the patient, a part of the tissue sample will be saved in order to carry out the analysis planned for the research.

INTERVENTIONS:
Other: During the surgery planned as part of the routine care of the patient, a part of the tissue sample will be saved in order to carry out the analysis planned for the research. — During the surgery planned as part of the routine care of the patient, a part of the tissue sample will be saved in order to carry out the analysis planned for the research.

SUMMARY:
Neuromuscular diseases (NMDs) affecting motor neurons (MN) induce progressive muscle denervation, and become fatal when respiratory muscles e.g. the diaphragm are affected and can no longer contract. In some cases, such as Charcot's disease (Amyotrophic lateral sclerosis-ALS), there is no cure and patients die due to respiratory failure few years after diagnosis. Investigations on NMD-induced alterations of respiratory muscles in humans are limited notably by the absence of available in vitro model based on cell cultures of diaphragm-derived myoblasts. Yet, this cell tool is likely to help in developing original therapies to limit diaphragm muscle atrophy and dysfunction in NMD. To date, only cell cultures of human myoblasts obtained from limb muscles are available, making difficult to transpose results to the diaphragm.

Thus, in the present project, we propose to :

1. originally develop primary cultures of myoblasts from human diaphragm, obtained from surgical resection of diaphragmatic endometriosis,
2. characterize them in terms of differentiation status (Histology, IF), metabolism (Metabolomics by NMR, cell respiration), and gene expression (RNASeq), in comparison to primary myoblasts cultures derived from the deltoid already available in the team.

This project will provide an original new tool and important data on the specificity of diaphragm-derived myoblasts, compared to limb muscle-derived myoblasts with the long-term perspective of opening new therapeutical pathways for patients with severe NMDs.

DETAILED DESCRIPTION:
Neuromuscular diseases (NMDs) affecting motor neurons (MN) induce progressive muscle denervation, and become fatal when respiratory muscles e.g. the diaphragm are affected and can no longer contract. In some cases, such as Charcot's disease (Amyotrophic lateral sclerosis-ALS), there is no cure and patients die due to respiratory failure few years after diagnosis. Investigations on NMD-induced alterations of respiratory muscles in humans are limited notably by the absence of available in vitro model based on cell cultures of diaphragm-derived myoblasts. Yet, this cell tool is likely to help in developing original therapies to limit diaphragm muscle atrophy and dysfunction in NMD. To date, only cell cultures of human myoblasts obtained from limb muscles are available, making difficult to transpose results to the diaphragm.

Thus, in the present project, we propose to :

1. originally develop primary cultures of myoblasts from human diaphragm, obtained from surgical resection of diaphragmatic endometriosis,
2. characterize them in terms of differentiation status (Histology, IF), metabolism (Metabolomics by NMR, cell respiration), and gene expression (RNASeq), in comparison to primary myoblasts cultures derived from the deltoid already available in the team.

This project will provide an original new tool and important data on the specificity of diaphragm-derived myoblasts, compared to limb muscle-derived myoblasts with the long-term perspective of opening new therapeutical pathways for patients with severe NMDs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* diaphragmatic endometriosis requiring surgical resection of the nodules in the diaphragm.
* Collection of non-opposition

Exclusion Criteria

* Inability to speak and/or read French
* Patients under tutor or curatorship
* Protected adults

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diaphragmatic endometriosis requiring surgical nodules resection in the diaphragm.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Molecular characteristics | Inclusion
  The primary endpoint will be the identification of molecular and cellular signatures specific of the diaphragm as compared with human deltoid muscle cultures, notably based on the study of :
  * differentiation, by studying the course of myoblast differentiation and fusion in polynucleated myotubes (IF Desmin, Slow and fast Myosin Heavy Chain),
  * energy metabolism (extra- and intra-cellular metabolomics by NMR, cell respiration by the Seahorse technology),
  * gene regulation, by analysing the transcriptomic signature (RNAseq).
Cellular characteristics | Inclusion
  The primary endpoint will be the identification of molecular and cellular signatures specific of the diaphragm as compared with human deltoid muscle cultures, notably based on the study of :
  * differentiation, by studying the course of myoblast differentiation and fusion in polynucleated myotubes (IF Desmin, Slow and fast Myosin Heavy Chain),
  * energy metabolism (extra- and intra-cellular metabolomics by NMR, cell respiration by the Seahorse technology),
  * gene regulation, by analysing the transcriptomic signature (RNAseq).

SECONDARY OUTCOMES:
Presence of diaphragm-derived myoblasts | Inclusion
  The secondary endpoint will be to build a library of molecular and cellular signatures for the major respiratory muscle i.e. the diaphragm in human. Decisive differences between cellular and molecular signatures across muscles (Diaphragm and Deltoid) will be analysed by principal component analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle NGUYEN, MD, PHD, Study Director — Physical Medicine and Rehabilitation Department - Cochin hospital; Marco ALIFANO, MD, PHD, Principal Investigator — Department of Thoracic Surgery - Cochin Hospital
Locations (1):
- Department of Thoracic Surgery - Cochin Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided